CLINICAL TRIAL: NCT04773834
Title: A Randomized Control Trial to Study the Effects of Automated Physician Directed Messaging on Patient Engagement in a Digital Diabetes Prevention Program
Brief Title: Evaluation of an Automated Physician-Directed Messaging on Patient Engagement in the Digital Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-01548; 1R18DK118545-01A1 (NIH)
Record Dates: First submitted 2020-12-29; First posted 2021-02-26 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will be enrolled virtually into a digital diabetes prevention program through the Noom app and willing to receive text messages based on their engagement levels in Noom from the study team, as well as complete text-based surveys.
  Interventions: Other: Digital diabetes prevention program (dDPP); Other: Adapted dDPP-EHR tool
- Control group (Other): Participants will be enrolled virtually into the digital diabetes prevention program through the Noom app and willing to receive general text messages from the study team
  Interventions: Other: Digital diabetes prevention program (dDPP)

INTERVENTIONS:
Other: Digital diabetes prevention program (dDPP) — The digital diabetes prevention program is through the Noom app, and the three devices (Fitbit physical activity tracker, Fitbit weight scale, and self-check hemoglobin a1c kit). This is a one year diabetes prevention program where participants will be expected to participate in 5 to 7 interviews over a 18 month period.
Other: Adapted dDPP-EHR tool — This is a product of Phase 1 and 2 of this study where participants will receive detailed text messaging regarding their engagement levels in Noom app.
  Arms: Experimental group

SUMMARY:
This study aims to understand the effects of automated physician directed messaging on patient engagement in the digital diabetes prevention program (dDPP). The messages are tailored to patient engagement levels based on established engagement thresholds, which are based on the patient's use of the dDPP application. The system is designed to minimize work for providers by sending automated targeted messages to patients to potentially increase engagement, prevent onset of diabetes and improve clinical outcomes. The patients in the study are automatically nudged using a combination of text messaging and MyChart messaging.

DETAILED DESCRIPTION:
Using a mixed-methods design, this study will be completed in three phases. For Phase 3, we aim to conduct a randomized control trial with 400 patients with pre-diabetic, all of whom will be using the dDPP application. Half of enrolled patients will be randomized to the intervention group and receive automated targeted messaging.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, BMI ≥ 25 kg/m2 (> 22 kg/m2 if self-identified as Asian)
* Must be a NYU Langone patient
* A diagnosis of prediabetes (either diagnosis of prediabetes or an HbA1C level of 5.7%-6.4% in past 12 months) or diabetes risk factors (BMI ≥ 25 kg/m2 or > 22 kg/m2 if self-identified as Asian
* Safe to engage in moderate physical exercise (as determined by their PCP)
* Sufficient English to be able to complete the enrollment process
* Has app-capable device with data to use the dDPP application and receive text messages

Exclusion Criteria:

* Diagnosed with diabetes
* Patients whose weight may vary considerably over the study's timeframe for reasons other than the intervention (e.g. cancer, pregnancy, ascites, severe CHF)
* Patients with severe psychiatric disease or dementia
* Active health condition that prevents them from engaging in moderate exercise

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devin Mann, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to hibrid.lab@nyulangone.org To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Rodriguez DV, Chen J, Viswanadham RVN, Lawrence K, Mann D. Leveraging Machine Learning to Develop Digital Engagement Phenotypes of Users in a Digital Diabetes Prevention Program: Evaluation Study. JMIR AI. 2024 Mar 1;3:e47122. doi: 10.2196/47122. PMID 38875579

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 354 | 197
Completed | 284 | 151
Not Completed | 70 | 46
Not completed — UPID not claimed | 29 | 5
Not completed — Failed criteria for randomization | 41 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 284 | 151 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.2) | 57.4 (11.2) | 57.5 (11.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 188 | 100 | 288
  Male | 83 | 48 | 131
  Other | 2 | 0 | 2
  Missing | 11 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 24 | 51
  Not Hispanic or Latino | 187 | 95 | 282
  Unknown or Not Reported | 70 | 32 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 19 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 33 | 104
  White | 137 | 80 | 217
  More than one race | 34 | 16 | 50
  Unknown or Not Reported | 11 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 284 | 151 | 435

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) Level (mmol/Mol)
Description: Repeated measurements of participant HbA1c will be taken via HbA1C home test kit and electronic health records. Data will be collected at discrete time points: 0 month (at enrollment), 6 months, 12 months (study completion). Changes were assessed relative to baseline.
Time Frame: Baseline, Month 6
Population: The number of participants included in this analysis reflects the use of multiple imputation to account for missing data. All available cases were incorporated into the imputed datasets, and estimates are based on pooled results across imputations.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 284 | 151
mmol/mol | 0.02 (0.034) | -0.03 (0.045)

2. Primary Outcome: Change in Hemoglobin A1c (HbA1c) Level (mmol/Mol)
Description: as for outcome 1
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 284 | 151
mmol/mol | 0.01 (0.040) | 0.01 (0.043)

3. Primary Outcome: Change in Body Weight (Lbs)
Description: Repeated measurements of participant weight will be taken via remote Bluetooth-connected weight scales, measured in light clothing without shoes. Data will be collected at discrete time points: 0 month (at enrollment), 3 months, 6 months, 9 months, 12 months (study completion). Changes were assessed relative to baseline.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 284 | 151
lbs | -7.13 (0.968) | -7.02 (1.200)

4. Primary Outcome: Change in Body Weight (Lbs)
Description: as for outcome 3
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 284 | 151
lbs | -7.42 (0.993) | -7.02 (1.330)

5. Primary Outcome: Change in Body Mass Index (BMI) (Lbs/in^2)
Description: BMI was calculated using height (in) from electronic health records and weight (lbs) from remote Bluetooth-connected weight scales. Data was collected at discrete time points: 0 month (at enrollment), 3 months, 6 months, 9 months, 12 months (study completion). Changes were assessed relative to baseline.
Time Frame: Baseline, Month 6
Population: Only 163 participants in the experimental group and 94 participants in the control group were analyzed. The others were missing weight data at either 6 or 12 months and were excluded. This analysis was done separately from the other outcomes, which used multiple imputation to help fill in the missing data.
Measure: Mean (Standard Deviation); unit: lbs/in^2
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 163 | 94
lbs/in^2 | -1.1792 (0.150) | -1.30 (0.228)

6. Primary Outcome: Change in Body Mass Index (BMI) (Lbs/in^2)
Description: as for outcome 5
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: lbs/in^2
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 163 | 94
lbs/in^2 | 1.2045 (0.147) | -1.16 (0.218)

7. Secondary Outcome: Engagement With the dDPP Platform
Description: Engagement was defined as completion of the following Noom activities: submission of at least one weigh-in; reading one article per week; participation in socialization through either one group post per week or one message to a Noom coach; and meeting physical activity goals by achieving either 150 minutes of activity or the step target assigned by Noom. Outcome measure is assessed as as score on a scale, where 0=Fail, and 1=pass
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 284 | 151
score on a scale | 0.25 (0.0206) | 0.15 (0.029)

8. Secondary Outcome: Engagement With the dDPP Platform
Description: as for outcome 7
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 284 | 151
score on a scale | 0.29 (0.048) | 0.25 (0.061)

ADVERSE EVENTS:
Time Frame: SAEs and AEs were assessed until the end of treatment.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/151
Other Adverse Events (participants affected / at risk) | 0/284 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT04773834/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04773834/ICF_000.pdf